CLINICAL TRIAL: NCT06489145
Title: Users' Experience and Cognitive Improvement in High-technology Rehabilitation Programs for Post-stroke Patients: a Multi-method, Multi-informant, Patient-centred Approach
Brief Title: Multi-domain Improvements in High-TEchnology Rehabilitation Programs for Post-stroke Patients
Acronym: ITER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milano Bicocca (Other)
Collaborators: University of Milan (Other); Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Principal Investigator, Marco D'Addario, Associate Professor, University of Milano Bicocca
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0025654/24; RM-2024-803 (Other: University of Milano-Bicocca)
Record Dates: First submitted 2024-06-25; First posted 2024-07-05 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-07

CONDITIONS: Stroke
Keywords: Stroke Rehabilitation; Technology; Cognition; Quality of Life; Well-Being; Experience of Use
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Technology-enhanced Rehabilitation (Experimental): Patients will participate in technology-enhanced rehabilitation programs in addition to multidisciplinary traditional treatment.
  Interventions: Device: Technology-enhanced Rehabilitation; Other: Multidisciplinary Traditional Rehabiltiation
- Standard Rehabilitation (Active Comparator): Patients will participate in multidisciplinary traditional treatment only
  Interventions: Other: Multidisciplinary Traditional Rehabiltiation

INTERVENTIONS:
Device: Technology-enhanced Rehabilitation — Based on their individualized rehabilitation project, patients will undergo robot-assisted therapy (RAT) and/or virtual reality (VR)-based treatment.
  RAT will consist of the use exoskeleton devices intended for the treatment of upper limbs (Armeo-Spring™) or for the lower limbs (Lokomat™) impairments.
  VR-based rehabilitation will be conducted non-immersive VR devices: the ProKin 252™ (TechnoBody SRL, Italy), the D-Wall™ (TechnoBody SRL, Italy), and the Walker View™ (TechnoBody SRL, Italy).
  Technology-enhanced treatment duration (number of sessions, minutes of use) will strictly depend on patients' rehabilitation needs and individualized rehabilitation program. Overall, part of the duration of the whole treatment will be dedicated to the use of the technological device, resulting in the same amount of rehabilitation for all participants.
  Arms: Technology-enhanced Rehabilitation
Other: Multidisciplinary Traditional Rehabiltiation — Patients will receive traditional treatment consisting of two daily one-hour session (4 weeks, 20 sessions) and including rehabilitation activities like range of motion exercises (passive, active assisted and active), progressive resistive exercises, balance and strength training, and aerobic conditioning. The intervention procedures will follow the routine multidisciplinary clinical practice of the Institute where the study will be carried out. Procedures will be adapted according to patient's medical diagnosis, disability severity, and to the consequent rehabilitation objectives in favor of an individualized rehabilitation project and program. If necessary, patients might therefore undergo parallel rehabilitation activities (ie, occupational therapy, speech therapy, cognitive stimulation) that will be kept under control throughout data collection and analyses.

SUMMARY:
Through a multi-method, multi-informant, and patient-centred approach, the study aims to investigate the experience of use and the effectiveness of rehabilitation technology (robotics and virtual reality - VR) in post-stroke patients and their caregivers and therapists

DETAILED DESCRIPTION:
The present research will consist of two parallel studies.

Study 1 (ID: 0025654/24). As a first goal the study aims to investigate pre- post-intervention changes on patients' motor, functional, cognitive, psychological and quality of life outcomes. Intervention effects will be estimated among patients participating in technology-enhanced rehabilitation programs and compared to those undergoing traditional treatment only.

As a second goal, the study aims to evaluate patients' subjective rehabilitation experience, treatment expectations and compliance, and (in case of technology use) devices usability, acceptability and psychosocial impact.

As a third goal, the study aims to extend the evaluation on rehabilitation experience to patients' caregivers, specifically investigating their treatment expectations and, at the end of the intervention, treatment satisfaction.

As a fourth goal, the study aims to evaluate the rehabilitation experience and technology experience of use in patients' therapists, specifically investigating their treatment expectations and, at the end of the intervention, patients' compliance and participation levels in the treatment.

Study 2 (ID: RM-2024-803). Therapists will be also involved in a parallel qualitative investigation through focus-groups to further explore the barriers and facilitators related to the implementation of technological devices into post-stroke rehabilitation programs.

ELIGIBILITY:
Study 1 (ID: 0025654/24)

Patients

Inclusion Criteria:

* Acute stroke event occurring within a maximum of 12 months prior to treatment;
* Age over 18 years;
* Acceptable hyposthenia evaluated with the Motricity Index (scores less than the maximum)
* Spasticity, if present, compatible with limb function (MAS score < 2)
* Mental health condition allowing for a full understanding of the study objectives and completion of self-report measures

Exclusion Criteria:

* Severe clinical condition (e.g., cognitive impairment - MMSE score < 24), presence of sever apraxia, complete upper limbs hemiplegia, severe upper limb sensory disorders, joint fractures and dislocations);
* clinical non-eligibility to the use of exoskeleton devices as per technical specifications of the devices
* Inability or difficulty in completing self-report measures in Italian and/or secondary illiteracy;
* Presence of psychiatric pathology in medical history or recent psychiatric pathology that could affect reliability of data collected;
* Refusal or withdrawal of informed consent at any stage of the study.

Caregivers

Inclusion Criteria:

* Any informal caregiver (e.g., family member, friend) who continuously assists the enrolled patient for at least half a day;

Exclusion Criteria:

* Inability or difficulty in understanding Italian language and/or illiteracy;
* Refusal or withdrawal of informed consent at any stage of the study

Therapists

Inclusion Criteria:

* Physiotherapists who assist enrolled patients throughout the entire intervention period

Exclusion Criteria:

* Physiotherapists who partially assist enrolled patients throughout the entire intervention period

Study 2 (ID: RM-2024-803)

Therapists

Inclusion Criteria:

* Physiotherapists who have sufficient professional experience in use of rehabilitation technology in post-stroke rehabilitation programs;

Exclusion Criteria:

* Refusal or withdrawal of informed consent at any stage of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Pre-post Intervention Change in Motor impairment | Baseline to 4-week follow-up
  Changes will be assessed with the Motricity Index (MI). Higher scores indicate lower motor impairment in terms of muscle strength and upper and lower limbs motricity (range: 0-33).
Pre-post Intervention Change in Spasticity | Baseline to 4-week follow-up
  Changes will be assessed with the Asworth modified Scale (MAS). Higher scores indicate higher spasticity (range: 0-4 for each body part assessed)
Pre-post Intervention Change in upper limbs sensory and motor functions | Baseline to 4-week follow-up
  Changes will be assessed with the Fugl-Meyer Upper Extremity Scale (FMUE). Higher scores indicate lower sensory-motor disability (Upper limb motor function, range: 0-66; lower limb motor function, range: 0-34; sensory function, range:0-24; balance, range: 0-14; joint range of motion, range: 0-44; joint pain, range:0-44).
Pre-post Intervention Change in Autonomy in Activities of Daily Living (ADLs) | Baseline to 4-week follow-up
  Changes will be assessed with the Barthel Index Modified (BIM). Higher scores (range: 0-100) indicate higher autonomy levels in ADLs (chair/bed transfer, ambulation, stair climbing, toilet transfer, bowel control, bladder control, bathing, dressing, personal hygiene, feeding).
Pre-post Intervention Change in Functional Disability | Baseline to 4-week follow-up
  Changes will be assessed with the Functional Independence Measure (FIM), which includes two sub-scales evaluating motor (range: 13-91) and cognitive (range: 5-35) domains in relation to disability. Higher scores indicate lower levels of motor and cognitive disability.
Pre-post Intervention Change in global cognition | Baseline to 4-week follow-up
  Changes will be assessed with the Mini Mental State Examination (MMSE), which includes sub-scores on temporal and spatial orientation, attention, executive functions, memory, language, and visual-spatial abilities. Higher scores indicate better global cognitive functioning (range: 0-30)
Pre-post Intervention Change in Long-term Verbal Memory | Baseline to 4-week follow-up
  Changes will assessed with the Rey Auditory Verbal Memory Test (RAVLT). Higher scores indicate better long-term verbal memory functioning (range: 0-15)
Pre-post Intervention Change in Short-term Verbal Memory | Baseline to 4-week follow-up
  Changes will be assessed with the Digit Span Task (DST). Higher scores indicate better short-term verbal memory functioning (range: 3-9)
Pre-post Intervention Change in Long-term Visual-spatial Memory | Baseline to 4-week follow-up
  Changes will be assessed with the Rey-Osterrieth Complex Figure Test. Higher scores indicate better long-term visual.spatial memory functioning (range: 0-36)
Pre-post Intervention Change in Short-term Visual-spatial Memory | Baseline to 4-week follow-up
  Changes will be assessed with the Corsi Block-Tapping Test. Higher scores indicate better short-term visual-spatial memory functioning (range: 3-9)
Pre-post Intervention Change in Visual-Spatial Attention | Baseline to 4-week follow-up
  Changes will be assessed with the Multiple Features Target Cancellation (MFTC) test. Higher scores indicate better attentional and visual search abilities (range: 0-13)
Pre-post Intervention Change in Executive Functions | Baseline to 4-week follow-up
  Changes will be assessed with the Trail Making Test (TMT). Higher time scores (i.e., seconds) indicate worse divided attention, cognitive flexibility, shifting and visual-motor coordination functions
Pre-post Intervention Change in Verbal Fluency | Baseline to 4-week follow-up
  Changes will be assessed with Phonemic and Semantic Verbal Fluency tests. Higher scores (i.e., number of words) indicated better linguistic and verbal fluency functions
Pre-post Intervention Change in Perceived Health Status | Baseline to 4-week follow-up
  Changes will be assessed with the EuroQoL Visual Analogue Scale (EQ-VAS). Higher scores indicate better perceived health status (range: 0-100)
Pre-post Intervention Change in Perceived Health-related Quality of Life | Baseline to 4-week follow-up
  Changes will be assessed with the Short-Form Health Survey-12 (SF-12). Higher scores in bot sub-scales (Mental Health and Physical Health) indicate better perceived health-related quality of life (range: 0-100)
Pre-post Intervention Change in Anxiety and Depression Symptoms | Baseline to 4-week follow-up
  Changes will be assessed with the Hospital Anxiety and Depression Scale (HADS). Higher scores indicated more severe anxiety and depression symptoms (range: 0-21)

SECONDARY OUTCOMES:
Change in Patient's Subjective Rehabilitation Experience | Baseline to 4-week follow-up (Repeated measures throughout the trial)
  Changes will be monitored through Ecological Momentary Assessment (EMA) method. Patients will be asked to fill out a daily diary after each therapy session and indicate their rehabilitation experience in terms of engagement, motivation, enjoyment and satisfaction. Selected items from the Intrinsic Motivation Inventory (IMI) will be administered. Higher scores indicate better subjective rehabilitation experience.
Rehabilitation Outcomes Expectations | Baseline
  Expectations will be assessed with the Expectancy sub-scale of the Credibility/Expectancy Questionnaire (CEQ). The assessment will be carried out on patients, their caregivers and therapists. Higher scores indicate more positive expectations on rehabilitation outcomes (range: 0-100)
Satisfaction with Rehabilitation Treatment | Baseline to 4-week follow-up
  Satisfaction levels in patients' caregivers will be assessed with Involvement practices scale. Higher scores indicate more positive caregiver's perception of information giving from rehabilitation staff, involvement in decision-making, and training to collaborate (range: 0-30)
Technology Perceived Usability | 4-week follow-up
  Perceived usability of the technological devices implemented will be assessed with the System Usability Scale (SUS). Higher scores indicate better technological device usability (range: 0-100)
Technology Acceptance | 4-week follow-up
  Acceptance will be assessed with the Technology Assisted Rehabilitation Patient Perception Questionnaire (TARPP-Q). Higher scores indicate higher technology acceptance in terms of engagement levels, usability, distress and perceived hindrance (range: 31-124)
Technology Psychosocial Impact | 4-week follow-up
  Psychosocial impact will be assessed with the Psychosocial Impact of Assistive Device Scale (PIADS). Higher scores indicate better impact on patient's perceived adaptability (range: -18/+18), ability (range: -36/+36), and self-esteem (range: -24/+24).

CONTACTS AND LOCATIONS:
Overall Officials: Patrizia Steca, PhD, Principal Investigator — University of Milano Bicocca; Marco D'Addario, PhD, Principal Investigator — University of Milano Bicocca; Alessandra Gorini, PhD, Principal Investigator — University of Milan
Locations (1):
- University of Milano-Bicocca, Milan, Italy